CLINICAL TRIAL: NCT01609140
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind Study of the Safety and Efficacy of MPSK3169A in Patients With Coronary Heart Disease or High Risk of Coronary Heart Disease
Brief Title: A Phase II Study of the Safety and Efficacy of MPSK3169A in Patients With Coronary Heart Disease or High Risk of Coronary Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC28210
Record Dates: First submitted 2012-05-24; First posted 2012-05-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Heart Disease
Keywords: Hyperlipidemia; Dyslipidemia
MeSH Terms: conditions — Coronary Disease; Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- A (Experimental)
  Interventions: Drug: MPSK3169A
- B (Experimental)
  Interventions: Drug: MPSK3169A
- C (Experimental)
  Interventions: Drug: MPSK3169A
- D (Experimental)
  Interventions: Drug: MPSK3169A
- E (Experimental)
  Interventions: Drug: MPSK3169A
- F (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MPSK3169A — Dose regimen A, repeating subcutaneous injections every 4 weeks
  Arms: A
Drug: MPSK3169A — Dose regimen E, repeating subcutaneous injections every 4 weeks
  Arms: E
Drug: MPSK3169A — Dose regimen D, repeating subcutaneous injections every 4 weeks
  Arms: D
Drug: MPSK3169A — Dose regimen C, repeating subcutaneous injections every 4 weeks
  Arms: C
Drug: MPSK3169A — Dose regimen B, repeating subcutaneous injections every 4 weeks
  Arms: B
Drug: Placebo — Repeating subcutaneous injections of placebo every 4 weeks
  Arms: F

SUMMARY:
The purpose of this study is to evaluate the safety and cholesterol lowering effects of MPSK3169A when given as subcutaneous (SC) injections over a 24-week period to patients with a high risk of cardiovascular events and LDL-c levels well above goal.

ELIGIBILITY:
Inclusion Criteria:

* Use of a standard-of-care statin at a stable dose, or intolerance of statins, without use of other lipid modifying therapies
* Fasting LDL cholesterol 90-250 mg/dL on the statin regimen above

And at least one of the following:

* Coronary heart disease (CHD) with a history of myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG), or prior coronary angiography demonstrating coronary atherosclerosis
* A CHD risk equivalent condition, including diabetes mellitus (type 1 or 2), chronic kidney disease, prior stroke, carotid disease, peripheral arterial disease, or abdominal aortic aneurism
* >/=2 CHD risk factors (age >/= 45 years for men or >/= 55 years for women; smoking; hypertension; low HDL cholesterol; family history of premature CHD) and a high risk of a CV event based on risk estimation systems

Exclusion Criteria:

* Severe congestive heart failure (NYHA Class III-IV) or left ventricular ejection fraction </= 35%
* Recent (within 3 months) MI, unstable angina, stroke, transient ischemic attack, CABG, PCI, hospital admission for heart failure, major surgery, uncontrolled cardiac arrhythmia (other than atrial fibrillation or flutter), or initiation of renal replacement therapy (dialysis)
* Fasting serum triglyceride level >/= 400 mg/dL
* Homozygous familial hypercholesterolemia
* Poorly controlled diabetes mellitus, hypertension or thyroid disease
* Liver or muscle disease, including abnormal test results at screening
* Pregnant or lactating

The above list is not intended to contain all factors relevant to a patient's eligibility for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in LDL-c concentration | at Day 169

SECONDARY OUTCOMES:
Absolute change from baseline in LDL-c concentration for each arm at the nadir for that arm | over the 24 week treatment period
Average value over time of the change in LDL-c (absolute and percent change) for each arm, up to Day 169, weighted by the number of weeks between consecutive LDL-c measurements | up to Day 169
Percent change from baseline in LDL-c concentration at Day 169 and at the nadir for each arm | at Day 169 and over the 24 week treatment period
Percent and absolute change from baseline in LDL-c concentration at all other designated timepoints | at all other designated timepoints
Percent and absolute change from baseline in total cholesterol, non-HDL-c, and apolipoprotein B (ApoB) at Day 169 and at the nadir for each arm | at Day 169 and over the 24 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (67):
- United States (32):
  - Goodyear, Arizona
  - Carmichael, California
  - Spring Valley, California
  - Walnut Creek, California
  - Wildomar, California
  - Jacksonville, Florida
  - Ponte Verde, Florida
  - Boise, Idaho
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Auburn, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - St Louis, Missouri
  - Rochester, New York
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Springdale, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Knoxville, Tennessee
  - Boerne, Texas
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Wenatchee, Washington
- Canada (9):
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Sarnia, Ontario
  - Toronto, Ontario
  - Woodstock, Ontario
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
  - Sainte-Foy, Quebec
  - Trois-Rivières, Quebec
- Czechia (5):
  - Hodonín
  - Jičícin
  - Mariánské Lázně
  - Ostrava - Poruba
  - Rakovník
- Germany (2):
  - Berlin
  - Cologne
- Hungary (4):
  - Komárom
  - Nagykanizsa
  - Nyíregyháza
  - Sopron
- New Zealand (4):
  - Auckland
  - Christchurch
  - Nelson
  - Tauranga
- Norway (4):
  - Elverum
  - Hamar
  - Oslo
  - Sandnes
- Slovakia (4):
  - Bardejov
  - Bratislava
  - Prešov
  - Rimavská Sobota
- South Africa (3):
  - Cape Town
  - Centurion
  - Pretoria

REFERENCES:
- [Derived] Baruch A, Mosesova S, Davis JD, Budha N, Vilimovskij A, Kahn R, Peng K, Cowan KJ, Harris LP, Gelzleichter T, Lehrer J, Davis JC Jr, Tingley WG. Effects of RG7652, a Monoclonal Antibody Against PCSK9, on LDL-C, LDL-C Subfractions, and Inflammatory Biomarkers in Patients at High Risk of or With Established Coronary Heart Disease (from the Phase 2 EQUATOR Study). Am J Cardiol. 2017 May 15;119(10):1576-1583. doi: 10.1016/j.amjcard.2017.02.020. Epub 2017 Mar 1. PMID 28343601